CLINICAL TRIAL: NCT06164236
Title: Study of Predictors of Failure of Sulprostone Treatment in Postpartum Hemorrhage
Acronym: NALAPOST
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8013
Record Dates: First submitted 2020-11-02; First posted 2023-12-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum haemorrhage; Maternal morbidity; Oxytocin; Sulprostone; Uterine Hemorrhage; Obstetric Labor Complications
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Hemorrhage; Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators wish to identify potential factors predicting failure of second-line drug treatment (sulproston (Nalador®)): risk factors and factors linked to a failure to take initial care for PPH.

A better understanding of the aggravating factors of HPP and more particularly the factors inherent to the initial care would make it possible to think of ways to improve practices.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject having given birth at HUS or CHU Poissy Saint-Germain-en Laye between 01/01/2019 and 31/12/2020
* Subject having presented a postpartum haemorrhage treated with Sulprostone
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult person (≥18 years old) who gave birth at HUS or at Poissy Saint-Germain-en Laye university hospital between 01/01/2019 and 12/31/2020 and having presented a postpartum hemorrhage treated with Sulprostone
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
This a rétrospective study trayning to identify a potential predictors of failure of second-line drug treatment in the case of severe postpartum hemorrhage | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- École de sages-femmes de Strasbourg, Strasbourg, Starsbourg, France

REFERENCES:
- [Derived] Voillequin S, Meyer MN, Faraci F, Rozenberg MP, Rousseau A. Maternal and clinical characteristics associated with sulprostone failure in postpartum haemorrhage after vaginal delivery: A retrospective cohort study. Eur J Obstet Gynecol Reprod Biol. 2026 Feb;317:114862. doi: 10.1016/j.ejogrb.2025.114862. Epub 2025 Nov 28. PMID 41319511